CLINICAL TRIAL: NCT07105904
Title: Biological and Clinical Relevance of Quantra Viscoelastic Hemostatic Assay in Hemorrhagic Cardiac Surgery: a Prospective Observational Study
Brief Title: Biological and Clinical Relevance of Quantra Viscoelastic Hemostatic Assay in Hemorrhagic Cardiac Surgery
Acronym: QASH
Status: Recruiting | Type: Observational
Sponsor: Pitié-Salpêtrière Hospital (Other)
Responsible Party: Principal Investigator, Marquet Yann, Medical Doctor, Pitié-Salpêtrière Hospital
Other Study IDs: IRB 00010254 - 2025 - 065
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hemorrhage; Cardiac Surgery; Hemorrhagic Shock
Keywords: hemmorhage; hemorrhagic cardiac surgery; Quantra; viscoelastometric assay; cardiac surgery
MeSH Terms: conditions — Hemorrhage; Shock, Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Monocentric consecutive patients undergoing cardiac surgery: Monocentric consecutive patients undergoing cardiac surgery, tested for biological hemostasis during surgery with both viscoelastometric assay (Quantra Qplus) and QT, ACT, fibrinogenemia, platelet count.
  Interventions: Diagnostic Test: Viscoelastometric hemostatic assay

INTERVENTIONS:
Diagnostic Test: Viscoelastometric hemostatic assay — As part of usual care, when weaning the patient from CPB during cardiac surgery, blood samples are withdrawn from the patient to assess hemostasis: we test both Quantra viscoelastometric assay and biological hemostasis including QT, ACT, fibrinogen and platelet count
  Other Names: Quantra

SUMMARY:
The goal of this observational study is to assess the correlation between Quantra viscoelastometric assay and laboratory hemostasis biology in a cardiac surgery cohort presenting with acute hemorrhage in the operating room. The main questions it aims to answer are:

* is Quantra a valuable surrogate for hemostasis biology in the setting of bleeding cardiac surgery?
* are Quantra parameters well correlated with tranfusion thresholds in the setting of bleeding cardiac surgery?

DETAILED DESCRIPTION:
This observational study aims to assess the relevance of Quantra use in the setting of cardiac surgery patients presenting with acute bleeding in the operating room.

Hemorrhage is frequent in cardiac surgery. In the setting of per-operative acute bleeding, patient management and transfusions require a meticulous approach as both under-treatment and over-treatment can concur to morbidity and mortality. In this specific setting, the short timeframe of management usually does not allow usual laboratory tests (prothrombin time, activated clotting time, fibrinogen and platelets counts) to be integrated in the decision-making process. Viscoelastic hemostatic assays (VHA) such as Quantra might be relevant in this setting, owing to point-of-care bedside features.

As part of usual care for patients undergoing cardiopulmonary bypass for cardiac surgery at the Pitié-Salpêtrière Hospital, the investigators use Quantra viscoelastometric tests in various situations , including for per-operative hemorrhage management. Yet, it appears Quantra relevance has never been challenged in this population.

The investigators seek to determine whether in a population of patients presenting with significant hemorrhage in the operating room of cardiac surgery Quantra parameters (CT, CTH, FCS and PCS) are well-correlated to standard biology testing (prothrombin time, activated clotting time, fibrinogen and platelets count) and to transfusion thresholds.

Universal Definition of Perioperative Bleeding (UDPB) is a widely used quantification of bleeding in cardiac surgery. Nonetheless, most of its parameters of interest are assessed post-operatively and definition of acute bleeding during cardiac surgery lack. The investigators propose a modified UDPB definition to properly match significant per-operative bleeding events. Three sub-groups of patients will be considered for statistical analyses: patients presenting with severe hemorrhage, patients presenting with massive hemorrhage, and the others.

Severe hemorrhage will be defined when one or more of the following occur:

* no sternal closure or use of a modified closure strategy (such as GoreTex closure)
* use of 5 to 10 blood products (packed red blood cells (RBC), fresh frozen plasma (FFP), platelets) during surgery
* more than 4.5g of fibrinogen cryoprecipitate or concentrate administered during surgery
* more than 50 UI/kg of human prothrombin complex (PPSB) administered during surgery
* three different hemostatic products within FFP, platelets, fibrinogen products and PPSB administered during surgery
* re-infusion of more than 1000mL of blood recovered from cell-salvage process

Massive hemorrhage will be defined as one or more of the following:

* use of more than 10 blood products (RBC, FFP, platelets) during surgery
* use of recombinant activated factor VII during surgery
* use of all hemostatic products available (FFP, platelets, PPSB, fibrinogen products).

This study is conducted in accordance with French law pending to observational studies. Non-opposition of patients is assessed prior to inclusion and data collection. Registry datas are extracted from the patients's medical records after anonymization.

Sample size has been estimated considering that 70 patients with acute bleeding in the operating room will be needed to properly assess correlation between Quantra and hemostasis biology in this population of interest. Considering a 15% incidence of bleeding in the hospital, 600 patients should be included overall to attain this objective. Yearly, 1200 to 1300 patients undergo cardiopulmonary bypass for cardiac surgery at the Pitié-Salpêtrière hospital. Quantra viscoelastometric assay and hemostasis biology are part of usual care and are usually tested when weaning cardiopulmonary bypass (i.e. after protamin antagonization) when risk factors for bleeding are present. Considering Quantra consumption from previous years (>1000/y in 2023 and 2024), although multiple testing is possible for some bleeding patients, the investigators estimate that about half of the patients are tested for both Quantra and hemostasis biology at the time of weaning from CPB. Hence, it is planned to include prospective patients undergoing cardiac surgery with CPB for 1 year.

Statistical analysis will be computed by the investigators. Results for categorical variables, expressed as number (%), will be compared using the χ² test or Fisher's exact test when appropriate. Continuous variables, expressed as mean (± standard deviation) or median [25th-75th percentile interquartile range (IQR)], will be compared using Student's t-test or Wilcoxon's rank-sum test, depending on data distribution. Missing datas will be excluded from statistical analysis. Correlations between Quantra parameters and Prothrombin Time, Activated Clotting Time, fibrinogen count and platelet counts will be analyzed by Spearman-Rank test. Statistical association between Quantra parameters and transfusion thresholds will be assessed by Receiver Operating Characteristics (ROC) curves and extraction of best thresholds with Youden points.

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgery with cardiopulmonary bypass
* adult patient

Exclusion Criteria:

* no hemostatic assay including Quantra during surgery
* no hemostatic assay including standard biology (PT, ACT, fibrinogen concentration and platelet count) during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Monocentric prospective population of consecutive patients undergoing cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-07-09 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Correlation of Quantra with Prothrombin Time and Activated Clotting Time in patients presenting with acute bleeding in the operating room | From enrollment to 1 month post-operatively
  In the subgroup of patients presenting with either severe or massive hemorrhage as defined previously: correlation between Clotting Time without or with Heparinase (CT / CTH) with Prothrombin Time (PT) and Activated Clotting Time (ACT), all measured in seconds
Correlation of Quantra with fibrinogen concentration in patients presenting with acute bleeding in the operating room | From enrollment to 1 month post-operatively
  In the subgroup of patients presenting with either severe or massive hemorrhage as defined previously: correlation between Fibrinogen contribution to Clot Stiffness (FCS), in hPa, and patient's blood fibrinogen concentration in g/L
Correlation of Quantra with platelet count in patients presenting with acute bleeding in the operating room | From enrollment to 1 month post-operatively
  In the subgroup of patients presenting with either severe or massive hemorrhage as defined previously: correlation between Platelet contribution to Clot Stiffness (PCS), in hPa, and patient's platelet count in G/L

SECONDARY OUTCOMES:
Correlation of Quantra with Prothrombin Time (PT) and Activated Clotting Time (ACT) in patients without bleeding | From enrollment to 1 month post-operatively
  In the subgroup of patients not presenting with acute bleeding in the operating room: correlation between Clotting Time without or with Heparinase (CT / CTH) with Prothrombin Time (PT) and Activated Clotting Time (ACT), all measured in seconds
Correlation of Quantra with fibrinogen concentration in patients without bleeding | From enrollment to 1 month post-operatively
  In the subgroup of patients not presenting with acute bleeding in the operating room: correlation between Fibrinogen contribution to Clot Stiffness (FCS), in hPa, and patient's blood fibrinogen concentration in g/L
Correlation of Quantra with platelet count in patients without bleeding | From enrollment to 1 month post-operatively
  In the subgroup of patients not presenting with acute bleeding in the operating room: correlation between Platelet contribution to Clot Stiffness (PCS), in hPa, and patient's platelet count in G/L
Correlation between Quantra and prothrombin time transfusion threshold in patients presenting with hemorrhage in cardiac surgery | From enrollment to 1 month post-operatively
  In the subgroup of patients presenting with either severe or massive hemorrhage as defined previously: correlation between Clotting Time without or with Heparinase (CT / CTH) and Prothrombin Time < 50%
Correlation between Quantra and fibrinogen concentration transfusion thresholds in patients presenting with hemorrhage in cardiac surgery | From enrollment to 1 month post-operatively
  In the subgroup of patients presenting with either severe or massive hemorrhage as defined previously: correlation between Fibrinogen contribution to Clot Stiffness (FCS), in hPa, and patient's blood fibrinogen concentration <1.5g/L
Correlation between Quantra and platelet count transfusion thresholds in patients presenting with hemorrhage in cardiac surgery | From enrollment to 1 month post-operatively
  In the subgroup of patients presenting with either severe or massive hemorrhage as defined previously: correlation between Platelet contribution to Clot Stiffness (PCS), in hPa, and patient's platelet count <50G/L

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Bouglé, Md, PhD, Study Director — Pitié-Salpêtrière Hospital; Geoffroy Hariri, MD, Study Chair — Pitié-Salpêtrière Hospital; Pierre Basse, MD, Study Chair — Pitié-Salpêtrière Hospital
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, ICF
Time Frame: From July 2025 to July 2027
Access Criteria: Contact to principal investigator who will then refer to the study sponsor (Assistance Publique-Hopitaux de Paris, Hôpital de la Pitié-Salpêtrière)

REFERENCES:
- [Background] Dyke C, Aronson S, Dietrich W, Hofmann A, Karkouti K, Levi M, Murphy GJ, Sellke FW, Shore-Lesserson L, von Heymann C, Ranucci M. Universal definition of perioperative bleeding in adult cardiac surgery. J Thorac Cardiovasc Surg. 2014 May;147(5):1458-1463.e1. doi: 10.1016/j.jtcvs.2013.10.070. Epub 2013 Dec 9. PMID 24332097
- [Background] Naik BI, Tanaka K, Sudhagoni RG, Viola F. Prediction of hypofibrinogenemia and thrombocytopenia at the point of care with the Quantra(R) QPlus(R) System. Thromb Res. 2021 Jan;197:88-93. doi: 10.1016/j.thromres.2020.11.008. Epub 2020 Nov 10. PMID 33197797
- [Background] Huffmyer JL, Fernandez LG, Haghighian C, Terkawi AS, Groves DS. Comparison of SEER Sonorheometry With Rotational Thromboelastometry and Laboratory Parameters in Cardiac Surgery. Anesth Analg. 2016 Dec;123(6):1390-1399. doi: 10.1213/ANE.0000000000001507. PMID 27749339
- [Background] Achneck HE, Sileshi B, Parikh A, Milano CA, Welsby IJ, Lawson JH. Pathophysiology of bleeding and clotting in the cardiac surgery patient: from vascular endothelium to circulatory assist device surface. Circulation. 2010 Nov 16;122(20):2068-77. doi: 10.1161/CIRCULATIONAHA.110.936773. No abstract available. PMID 21098468